CLINICAL TRIAL: NCT03640000
Title: Acute Changes in Bioimpedance During Cardia Resynchronization Therapy
Brief Title: Acute Changes in Bioimpedance During Cardiac Resynchronization Therapy
Acronym: Impel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Hans Henrik Odland, principal Investigator, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014/1223
Record Dates: First submitted 2016-10-30; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Heart Failure, Systolic
MeSH Terms: conditions — Heart Failure, Systolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Determination of impedance signals (Experimental): This single arm study is designed to measure impedance signals from implanted leads in different positions in the heart. Signals obtained at different pre specified position are compared to each other to determine the robustness of the acquired measurements.
  Interventions: Diagnostic Test: Impedance measurements in Cardiac Resynchronization therapy

INTERVENTIONS:
Diagnostic Test: Impedance measurements in Cardiac Resynchronization therapy — Bioimpedance measurements

SUMMARY:
This study aims at Optimizing measured parameters to reflect underlying pathology in dyssynchronous hearts. This is an experimental study in patients were bioimpedance measurements are performed during implantation.

DETAILED DESCRIPTION:
Patients who are eligible for implantation af a Cardiac Resynchronization Therapy Device according to European Society of Cardiology guidelines are included. Measurements are performed on implanted leads and stored for post Processing. The study entry ends for each patient With completion of the implantation procedure.

ELIGIBILITY:
- Indication for Cardiac resynchronization therapy or Upgrade of exciting Device according to the current European Society of Cardiology guidelines.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-01; Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Optimization of Bioimpedance measurements | 3 years
  Acquisition of absolute and imaginary bioimpedance signals from electrodes of known location within the heart at different input current frequencies. Pacing is performed from Three different electrodes during acquisition of bioimpedance acquisition forming Three different groups. Wavelets of the signals are analyzed within each Group and compared within the Group and between the Groups. Optimization is achived when a discrimination factor that is calculated is improved.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Henrik Odland, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No